CLINICAL TRIAL: NCT01327352
Title: A Single Center, Non-randomized, Placebo Controlled Study for the Evaluation of the Influence of Food Regimen on Oshadi D Absorption
Brief Title: Evaluation of the Influence of Food Regimen on Oshadi D Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OS-DN-P1b-01
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oshadi D (Experimental): 2 dose levels of Oshadi D in 2 food regimen will be administered as following:
  * Subjects will receive placebo on the morning of day 1 during fast. Late breakfast will be provided 4 hours following placebo administration.
  * On day 8 a single dose of 180mg Oshadi D will be administrated during fast. Late breakfast will be provided 4 hours following drug administration
  * On day 16 subjects will be administered with 360mg of Oshadi D during fast. Late breakfast will be provided 4 hours following drug administration.
  * On day 24, 180mg of Oshadi D will be administrated immediately after breakfast.
  * On day 32, subject will be administered with 360mg of Oshadi immediately after breakfast.
  Interventions: Drug: Oshadi D

INTERVENTIONS:
Drug: Oshadi D — oral administration

SUMMARY:
The study will be a non-randomized, open label, single dose, placebo control, single center, and single arm study in healthy subjects. The study will include one administration of placebo and four single administrations of Oshadi D in two different dose levels, administered in two feeding regimen for the evaluation of the influence of food on Oshadi D absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male/female 21 years old and up.
* Subject must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.
* Subject must be sterile or infertile or use an approved method of contraception from the time that the first dose of study medication is taken until three months following study completion or discontinuation.

Exclusion Criteria:

* Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Subject with positive HIV serology or positive HBsAg at screening.
* History or evidence of any active liver disease.
* Female subject who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Inability to give written informed consent
* History of alcohol or drug abuse within 6 months of screening.
* Subject who have a positive urine drug screen for substances of abuse (benzodiazepine, THC, opiates, amphetamines, cocaine) at the screening.
* Mental disorders.
* Subject with poor venous access
* Significant swallowing disorders
* Digestive disorders;
* Small bowel surgery;
* Mall absorption disorders.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
DNase activity level (Kunitz/mL) for 2 dose levels, and different food regimen | 24 hours

SECONDARY OUTCOMES:
Maximum plasma DNase concentration (ng/mL) in different food regimen and dose levels | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Keren Duanis, MD, Principal Investigator — Assaf Harofe Medical Center, Israel; Hanna Levy, Dr., Study Director — Oshadi Drug Administration
Locations (1):
- Assaf Harofe Medical Center,, Zrifin, Israel